CLINICAL TRIAL: NCT01538134
Title: Antiphospholipid Antibodies and Early Fetal Growth Restriction (<34 Weeks of Gestation). A Case Control Study.
Brief Title: Antiphospholipid Antibodies and Fetal Growth Restriction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research & Development, Saint Thomas Hospital, Panama
Other Study IDs: MHST2012-01B
Record Dates: First submitted 2012-02-19; First posted 2012-02-23 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Fetal Growth Restriction; Antiphospholipid Syndrome
Keywords: Antibodies, anticardiolipin; Antibodies, B2 Glycoprotein I; Lupus Anticoagulant; Fetal Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation; Antiphospholipid Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients with ultrasonographic diagnosis of fetal growth restriction.
- Control: Patients with normal pregnancies at term.

SUMMARY:
The Antiphospholipid Syndrome is an immune disease where the presence of antibodies directed against cell membrane phospholipids (antiphospholipid antibodies) can cause an hypercoagulable state that causes thrombosis and obstetric complications (miscarriages, stillbirths). Since 1999 the Sapporo Criteria for Antiphospholipid Syndrome diagnosis includes the development of fetal growth restriction (diagnosed postpartum), but this was done without solid evidence of a relation between the two or using the most common form of fetal growth restriction diagnosis (ultrasound). Our study will try to add information to this particular point.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24-34 weeks.
* Ultrasonographic evidence of fetal growth restriction

  * Abdominal circumference < 3rd percentile.
  * Doppler with increase of placental resistance.

Exclusion Criteria:

* Known antiphospholipid syndrome.
* Known presence of antiphospholipid antibodies.
* Patients with systemic lupus erythematosus.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients admitted for fetal growth restriction (cases) and normal patients in labor at term (controls).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-02 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Lupus anticoagulant | 8 months
  Number of cases positive for Lupus Anticoagulant.
Anticardiolipin antibodies | 10 months
  Number of cases with high/medium levels of IgG/IgM of anticardiolipin antibodies.
B2 Glycoprotein I | 10 months
  Number of cases with levels of B2 Glycoprotein I > 99%

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Provincia de Panamá, Panama